CLINICAL TRIAL: NCT05681520
Title: Pilot of Peers Enhancing Engagement for Pain Services
Acronym: PEEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D4381-P; I21RX004381-01A1 (NIH)
Record Dates: First submitted 2022-12-16; First posted 2023-01-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; peer support
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single arm pilot study; intervention includes six 30-minute sessions with a peer specialist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- peer specialist (Experimental): Work with a peer specialist for six 30-minute sessions
  Interventions: Behavioral: PEEPS

INTERVENTIONS:
Behavioral: PEEPS — Working with a peer specialist for six 30-minute sessions to enhance engagement in pain management approaches/treatments
  Other Names: Peer Specialist Intervention

SUMMARY:
Chronic non-cancer pain is common among Veterans, and more work is needed to understand how best to support Veterans with chronic pain to improve pain-related function and quality of life. Peer specialists may be valuable resource to support Veterans in pain management. Peer specialists, individuals with lived experience who are hired and trained to work with Veterans, are increasingly being used outside traditional mental health settings. More research is needed to understand how best to train peer specialists to work in new settings and with new presenting problems, such as chronic pain. Peer support to help Veterans improve pain-related function, increase physical activity, and engage in recommended pain care, is especially needed. In this study, the investigators will finalize a peer-led intervention and then pilot it with 24 Veterans with chronic pain in order to establish feasibility and acceptability; results will be used to develop a larger proposal testing the intervention in a randomized trial.

DETAILED DESCRIPTION:
Background: Chronic pain, and particularly high-impact chronic pain (that is, pain last three months or longer that impacts daily functioning in one or more domains) is a leading cause of disability, often associated with declining functioning, lost days of work, and worsened quality of life. The Veterans Health Administration (VHA) identified both improved pain management and reduced opioid-related harms as national priorities, with an emphasis on improving function and pain-related disability. Peer specialists may be an untapped and valuable resource to support Veterans with chronic pain and enhance the effectiveness of pain treatment. Peer specialists are individuals with lived experience who work with Veterans to encourage patient activation and help patients manage chronic conditions. Peer specialists work in a variety of clinical settings, most commonly mental health clinics, and are well-suited to help patients who are harder to engage in services or those needing more support to promote self-management strategies. Peer support is particularly effective for patients with more severe illnesses or higher levels of distress, and thus may be helpful for Veterans with high-impact chronic pain.

Significance: Chronic pain is one of the most common and costly problems among Veterans using VHA healthcare. VHA guidelines for pain management and opioid therapy encourage non-pharmacological pain management strategies (NPMs) and non-opioid medications for chronic pain management. However, NPMs that emphasize improved pain-related function are often underutilized. Addressing pain management and opioid misuse are VHA priorities and this research directly aligns with VHA Rehabilitation Research & Development (RR&D) priorities, including promotion of non-pharmacological activity-based interventions for chronic pain, impacting outcomes such as pain; it also aligns with RR&D's broader goal of maximizing Veteran's function and quality of life.

Innovation & Impact: The role of peer specialists in VHA is rapidly expanding beyond traditional mental health settings, leading to an urgent need for additional research to understand how best to use peer specialists' unique skills to enhance care for Veterans in a wider range of settings. No studies to date have evaluated the use of peer specialists to support improvements in pain-related function among Veterans with chronic pain. The current proposal is innovative because it proposes, for the first time, using peer specialists to focus on pain management. If proven effective, this project could pave the way for widespread implementation of peer specialists into new settings where they can support pain management.

Specific Aims: The specific aims of this project are to (1) Use intervention mapping (IM) to refine the intervention, Peers Enhancing Engagement for Pain Services (PEEPS) and (2) Pilot test the feasibility and acceptability of PEEPS and collect function-focused outcome measures for use in a rigorous prospective study.

Methodology: After refining the intervention protocol using intervention mapping, the investigators propose a single arm pilot trial where the investigators will enroll 24 Veterans with high-impact chronic pain to participate in PEEPS, collecting data at baseline and three-months post baseline. The primary focus will be feasibility and acceptability; the investigators will also collect data on pain-related function, activity (steps walked, using pedometers), and well-being/quality of life.

Next Steps/Implementation: These data will inform the development of a larger proposal testing PEEPS in a multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Veteran receiving care from VA Connecticut Healthcare System
* referred to a VA Connecticut Pain Management Team
* has high-impact chronic pain as defined by the Graded Chronic Pain Scale - Revised
* willing/able to participate in sessions either in person or via video

Exclusion Criteria:

* moderate to severe cognitive impairment or apparent difficulty communicating with the research staff
* inability to read or understand English
* severely impaired hearing or speech that would preclude them from participating in telephone interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility - Number of completers | through study completion, approximately 18 months
  Number of Veterans who completed at least 3 sessions with the peer specialist
Acceptability | 3 months
  Intervention acceptability as indicated by results of qualitative interviews

SECONDARY OUTCOMES:
Feasibility - Recruiting 24 participants | through study completion, approximately 18 months
  Ability to recruit 24 participants over the study period
Feasibility - Enrollment of >15% of those invited | through study completion, approximately 18 months
  An enrollment rate of greater or equal to 15% of those invited to participate
Feasibility - Retention >60% | through study completion, approximately 18 months
  A retention rate of greater or equal to 60% of enrolled Veterans completing follow-up measures
Acceptability - Quantitative | 3 months
  Intervention acceptability as indicated by a score of 24 or greater on the CSQ-8

OTHER OUTCOMES:
Pain Interference | 3 months
  Brief Pain Inventory (BPI); we are piloting this measure for use in a future randomized trial. One-point decrease is often considered clinically meaningfully (range 0-10, lower scores are better).
Physical Function | 3 months
  Steps per day as measured by pedometer; we are piloting this measure for use in a future randomized trial. Improvement indicated by increased average steps per day.
Well-being | 3 months
  Well-Being Signs tool; we are piloting this three-item measure for use in a future randomized trial (higher scores are better, range 0-10)
Quality of Life | 3 months
  Health-related quality of life as measured by SF12; we are piloting this measure for use in a future randomized trial (range 0-100, higher scores are better)
Pain self-management | 3 months
  Modified version of Chronic Pain Coping Inventory (CPCI); we are piloting this measure for use in a future randomized trial. Improvement indicated by increased use of adaptive pain coping skills (items are scored 0 to 7, higher scores better)
Healthcare engagement | 3 months
  Altarum Consumer Engagement (ACE); we are piloting this measure for use in a future randomized trial. Improvement indicated by more engagement with healthcare (items are scored 1 to 5, high scores better)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Edmond, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication by contacting the study PI. Prior to distribution, a local privacy officer will certify that all datasets contains no PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available within 1 year of publication. The analytical datasets and statistical code used in the publication will be retained for 6 years, in accordance with VA record retention policy.
Access Criteria: Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement. De-identified data will be provided after requesters sign a Letter of Agreement detailing the mechanisms by which the data will be kept secure and access restricted to their study team and will state that the recipient will not attempt to identify any individual whose data are included and will not share the data.

DOCUMENTS (1):
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT05681520/ICF_000.pdf